CLINICAL TRIAL: NCT02319239
Title: Development of Prostate Cancer Stereotactic Radiotherapy in Tampere Using Intra-fractional Movement Detector and Diffusion-weighted Magnetic Resonance Imaging.
Brief Title: Prostate Cancer Stereotactic Radiotherapy
Acronym: ESKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETL R14009; R14009 (Other: TampereUH)
Record Dates: First submitted 2014-05-21; First posted 2014-12-18 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Prostate Neoplasms; Toxicity Due to Radiotherapy
Keywords: Prostate neoplasms; Urogenital neoplasms; Genital neoplasms, male; Radiation therapy; Prostate specific antigen; DW-MRI, diffusion weighted MRI; Intra-fractional movement; Hypofractionated radiotherapy; Stereotactic; Toxicity due to radiotherapy; Quality of life
MeSH Terms: conditions — Prostatic Neoplasms; Urogenital Neoplasms; Genital Neoplasms, Male | interventions — Chemical Fractionation; Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional fractionation (Active Comparator): During a radiotherapy period the prostate movement will be monitored by temporary implanted electromagnetic detector. Rectum fixation at 15/39 fractions. DW-MRI at baseline, 3 months and 12 months.
  Interventions: Radiation: Fractionation
- hypofractionated (Experimental): During a radiotherapy period the prostate movement will be monitored by temporary implanted electromagnetic detector. Rectum fixation at 10/20 fractions. DW-MRI at baseline, 3 months and 12 months.
  Interventions: Radiation: hypofractionated
- Stereotactic fractionation (Experimental): During a radiotherapy period the prostate movement will be monitored by temporary implanted electromagnetic detector. Rectum fixation at 5/5 fractions. DW-MRI at baseline, 3 months and 12 months.
  Interventions: Radiation: stereotactic fractionation

INTERVENTIONS:
Radiation: Fractionation — During a radiotherapy period the prostate movement will be monitored by temporary implanted electromagnetic detector. Rectum fixation at 15/39 fractions. DW-MRI at baseline, 3 months and 12 months.
  Arms: Conventional fractionation
Radiation: hypofractionated — During a radiotherapy period the prostate movement will be monitored by temporary implanted electromagnetic detector. Rectum fixation at 10/20 fractions. DW-MRI at baseline, 3 months and 12 months
  Arms: hypofractionated
Radiation: stereotactic fractionation — During a radiotherapy period the prostate movement will be monitored by temporary implanted electromagnetic detector. Rectum fixation at 5/5 fractions. DW-MRI at baseline, 3 months and 12 months
  Arms: Stereotactic fractionation

SUMMARY:
Primary purpose of the study is to develop a stereotactic radiation treatment (RT) to prostate cancer which minimizes treatment related toxicity. Movement of the prostate during a radiation therapy will be monitored by temporary implanted electromagnetic transmitter. This data will be used to define prostate marginals (PTV) for stereotactic treatment. Radiation toxicity to rectum will be reduced by using a rectum fixation during a treatment.

Study group I (20 patients) will be treated 39 x 2 Gy and study group II (20 patients) with 20 x 3 Gy fractionation schedules. With the data collected from these groups treatment marginals to prostate will be defined and used to treat group III (40 patients) with 5 x 7.25 Gy.

Second purpose of this study is to assess if Diffusion-weighted magnetic resonance imaging could be used to evaluate radiation treatment response in intermediate prostate cancer. Androgen deprivation therapy is not allowed in this study.

DETAILED DESCRIPTION:
New local prostate cancer patients needing external radiotherapy are included into three radiation dose groups;

Group I will be treated normal dosing (39 x 2 Gy) and study group II with hypofractionated dosing (20 x 3 Gy) and group III extreme hypofractionated dosing. Primary goal is to develop safe and effective curative radiotherapy for these patients

Second aim is to study Diffusion-weighted magnetic resonance image (DW MRI) in radiation treatment response in intermediate prostate cancer.

Patients are followed by MRI, PSA, bone scans and quality of life questionaries.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven prostate Cancer
* One or two risk factors for intermediate prostate cancer:

  * Gleason score 7
  * T2b-T2c
  * PSA 10-20 microg/l
* No need for androgen deprivation therapy
* Eligible fo MRI
* Radical radiotherapy

Exclusion Criteria:

* Locally advanced or metastatic prostate cancer
* Previous radiotherapy to pelvic reason
* Other severe disease
* Previous cancer within 5 years
* Severe urinary symptoms at the start of the study (over 20)
* Wide cavity after transurethral resection of prostate (TURP)

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
To determine whether the temporary implanted electromagnetic transmitter could be used to reduce treatment marginals in prostate cancer radiation therapy | 1 to 3 months
  Prostate specific antigen (PSA) recurrence

SECONDARY OUTCOMES:
Evaluation of DW-MRI to predict the outcome of prostate cancer radiation therapy | 0 - 12 months
  PSA recurrence
quality of life changes | 1 to 3 months
  questionaires

CONTACTS AND LOCATIONS:
Overall Officials: Petri Reinikainen, Principal Investigator — Tampere Unviersity Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Vanhanen A, Reinikainen P, Kapanen M. Radiation-induced prostate swelling during SBRT of the prostate. Acta Oncol. 2022 Jun;61(6):698-704. doi: 10.1080/0284186X.2022.2062682. Epub 2022 Apr 17. PMID 35435111
- [Derived] Vanhanen A, Poulsen P, Kapanen M. Dosimetric effect of intrafraction motion and different localization strategies in prostate SBRT. Phys Med. 2020 Jul;75:58-68. doi: 10.1016/j.ejmp.2020.06.010. Epub 2020 Jun 12. PMID 32540647
- [Derived] Vanhanen A, Syren H, Kapanen M. Localization accuracy of two electromagnetic tracking systems in prostate cancer radiotherapy: A comparison with fiducial marker based kilovoltage imaging. Phys Med. 2018 Dec;56:10-18. doi: 10.1016/j.ejmp.2018.11.007. Epub 2018 Nov 16. PMID 30527084